CLINICAL TRIAL: NCT04158479
Title: China Extracorporeal Life Support Registry
Status: Recruiting | Type: Observational
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Xiaotong Hou, Chief, Center for Cardiac Intensive Care, Beijing Anzhen Hospital
Other Study IDs: 2019040X
Record Dates: First submitted 2019-11-07; First posted 2019-11-08 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Cardiogenic Shock; Cardiac Arrest; Heart Failure; Acute Respiratory Distress Syndrome; Acute Respiratory Failure
MeSH Terms: conditions — Shock, Cardiogenic; Heart Arrest; Heart Failure; Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Pulmonary Support: ECMO support for acute respiratory failure, ARDS
  Interventions: Device: ECMO
- Cardiac Support: ECMO support for heart failure, cardiogenic shock
  Interventions: Device: ECMO
- Extracorporeal Cardiopulmonary Resuscitation: ECMO support for cardia arrest
  Interventions: Device: ECMO

INTERVENTIONS:
Device: ECMO — ECMO for circulatory and/or respiratory support

SUMMARY:
Extracorporeal life support (ECLS), also known as extracorporeal membrane oxygenation (ECMO), is an extracorporeal technique of providing effective cardiac and respiratory support to patients with lungs and/or heart failure. There was a growth in ECLS cases, centers, and center scale in China during the past decade.

This multi-center registry was conducted by Chinese Society of Extracorporeal Life Support. The objectives were to investigate China statistics of ECLS and to evaluate the short-term and long-term outcomes of patients with ECLS.

DETAILED DESCRIPTION:
Extracorporeal life support (ECLS), also known as extracorporeal membrane oxygenation (ECMO), is an extracorporeal technique of providing effective cardiac and respiratory support to patients with lungs and/or heart failure. There was a growth in ECLS cases, centers, and center scale in China during the past decade.

The objectives were to investigate China statistics of ECLS and to evaluate the short-term and long-term outcomes of patients with ECLS.

This multi-center registry was conducted by Chinese Society of Extracorporeal Life Support. Data were submitted by the following member institutions:

AFFILIATED HOSPITAL OF GUANGDONG MEDICAL UNIVERSITY, AFFILIATED HOSPITAL OF JINING MEDICAL UNIVERSITY, AFFILIATED HOSPITAL OF NANTONE UNIVERSITY, AFFILIATED HOSPITAL OF ZUNYI MEDICAL UNIVERSITY, ANHUI PROVINCIAL HOSPITAL, BEIJING ANZHEN HOSPITAL, CAPITAL MEDICAL UNIVERSITY, BEIJING CHILDREN'S HOSPITAL, CAPITAL MEDICAL UNIVERSITY, BEIJING FRIENDSHIP HOSPITAL, CAPITAL MEDICAL UNIVERSITY, BEIJING CHAO-YANG HOSPITAL, CAPITAL MEDICAL UNIVERSITY, BINZHOU MEDICAL UNIVERSITY HOSPITAL, CHANGHAI HOSPITAL, CHILDREN'S HOSPITAL OF SHANGHAI JIAOTONG UNIVERSITY, CHINESE PLA GENERAL HOSPITAL, DALIAN CENTRAL HOSPITAL, DONGGUAN PEOPLE'S HOSPITAL, FIRST AFFILIATED HOSPITAL OF KUNMING MEDICAL UNIVERSITY, FUJIAN PROVINCIAL HOSPITAL, FUZHOU PULMONARY HOSPITAL OF FUJIAN, GENERAL HOSPITAL OF NINGXIA MEDICAL UNIVERSITY, GUANGDONG PROVINCIAL PEOPLES HOSPITAL, HAINAN GENERAL HOSPITAL, HENAN PROVINCIAL CHEST HOSPITAL, HENAN PROVINCIAL PEOPLES HOSPITAL, NINGBO FIRST HOSPITAL (NINGBO HOSPITAL OF ZHEJIANG UNIVERSITY, PEKING UNION MEDICAL COLLEGE HOSPITAL, PEKING UNIVERSITY PEOPLE'S HOSPITAL, PEKING UNIVERSITY THIRD HOSPITAL, SHANXI PROVINCIAL PEOPLE'S HOSPITAL, SHENGJING HOSPITAL OF CHINAMESICAL UNIVERSITY, SHUNDE HOSPITAL OF SOUTHERN MEDICAL UNIVERSITY, SUZHOU MUNICIPAL HOSPITAL, TAIZHOU HOSPITAL OF ZHEJIANG PROVINCE, THE 2ND AFFILIATED HOSPITAL OF HARBIN MEDICAL UNIVERSITY, THE AFFILIATED HOSPITAL OF HANGZHOU NORMAL UNIVERSITY, THE AFFILIATED HOSPITAL OF QINGDAO UNIVERSITY, THE AFFILIATED HOSPITAL OF XUZHOU MEDICAL UNIVERSITY, THE CHILDREN'S HOSPITAL ZHEJIANG UNIVERSITY SCHOOL OF MEDICINE, THE FIRST AFFILIATED HOSPITAL OF ZHENGZHOU UNIVERSITY, THE FIRST AFFILIATED HOSPITAL OF CHONGQING MEDICAL UNIVERSITY, THE FIRST AFFILIATED HOSPITAL OF XIAMEN UNIVERSITY, THE FIRST AFFILIATED HOSPITAL WITH NANJING MEDICAL UNIVESITY, THE FIRST HOSPITAL AFFILIATED TO AMU (SOUTHWEST HOSPITAL), THE FIRST HOSPITAL OF LANZHOU UNIVERSITY, THE FIRST HOSPITAL OF ZHEJIANG PROVINCE, THE FIRST PEOPLE'S HOSPITAL OF YUEYANG, THE NORTHERN JIANGSU PEOPLES HOSPITAL, THE PEOPLE'S HOSPITAL OF GUANGXI ZHUANG AUTONOMOUS REGION, THE SECOND AFFILIATED HOSPITAL OF GUANGXI MEDICAL UNIVERSITY, THE SECOND AFFILIATED HOSPITAL OF ZHENGZHOU UNIVERSITY, THE SECOND AFFILIATED HOSPITAL OF ZHEJIANG UNIVERSITY SCHOOL OF MEDICINE, THE SECOND HOSPITAL OF JILIN UNIVERSITY, THE SECOND XIANGYA HOSPITAL OF CENTRAL SOUTH UNIVERSITY, THE SIXTH MEDICAL CENTER OF PLA GENERAL HOSPITAL, THE THIND AFFILIATED HOSPITAL OF XINJIANG MEDICAL UNIVERSITY, WEST CHINA HOSPITAL，SICHUAN UNIVERSITY, WUHAN ASIA HEART HOSPITAL, WUHAN JINYINTAN HOSPITAL, WUHAN UNION HOSPITAL, XIANGYIA HOSPITAL CENTRAL SOUTH UNIVERSITY, XIJING HOSPITAL, ZHEJIANG PROVINCE PEOPLE'S HOSPITAL, ZHON GNAN HOSPITAL OF WUHAN UNIVERSITY, ZHONGDA HOSPITAL SOUTHEAST UNIVERSITY, ZHONGSHAN HOSPITAL

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving ECMO for circulatory and/or respiratory support

Exclusion Criteria:

* Refusal of consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients receiving ECMO for circulatory and/or respiratory support
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 30 days

SECONDARY OUTCOMES:
All-cause mortality | 365 days
Rate of successful weaning from ECMO | 30 days
ECMO-related complications | 30 days
  Bleeding requiring transfusion or surgery, stroke, sepsis, limb ischemia requiring intervention, system or cannula change
Other complications | 30 days
  Acute renal failure, ulcer bleeding, pneumonia, sepsis
Duration stay at ICU and hospital | 365 days

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Cardiac Intensive Care, Beijing Anzhen Hospital, Capital Medical University, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Yuan Z, Liu Y, Wei G, Wang F, Yao B, Hou X, Xing J. Clinical characteristics of extracorporeal cardiopulmonary resuscitation in China: a multicenter retrospective study. BMC Anesthesiol. 2024 Jul 10;24(1):230. doi: 10.1186/s12871-024-02618-2. PMID 38987696